CLINICAL TRIAL: NCT04872543
Title: A Phase II Study of ASTX727 in Patients With PRC2 Loss Malignant Peripheral Nerve Sheath Tumor (MPNST)
Brief Title: A Study of ASTX727 in People With Malignant Peripheral Nerve Sheath Tumors (MPNST)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Taiho Pharmaceuticals, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-048; 1R01FD007544-01 (FDA); Philanthropy (Other: Philanthropy)
Record Dates: First submitted 2021-04-30; First posted 2021-05-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Malignant Peripheral Nerve Sheath Tumors (MPNST)
Keywords: ASTX727; Cedazuridine; Decitabine; PRC2 mutation; 21-048
MeSH Terms: conditions — Neurofibrosarcoma | interventions — decitabine and cedazuridine drug combination

STUDY DESIGN:
Intervention Model Description: This is a phase II trial to evaluate the efficacy of ASTX727 in patients with PRC2-loss MPNST.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ASTX727 (cedazuridine and decitabine) (Experimental): Patients who meet the eligibility criteria will be treated with oral ASTX727 (INQOVI) on days 1-5 of each 21-day cycle with Pegfilgrastim support on day 7. A delay in the start of subsequent cycles due to holidays, weather, or other circumstances will be permitted up to 7 days and not considered a protocol deviation. Drug dosing will be interrupted for any Grade 4 adverse events or clinically significant laboratory abnormalities. For Grade 3 or 4 AE, if the AE returns to Grade 1 or baseline, the patient may be re-escalated.
  Interventions: Drug: ASTX727

INTERVENTIONS:
Drug: ASTX727 — ASTX727 will be self-administered orally by the patient on a once daily basis, days 1 through 5 of each 21-day cycle. Cycle 1 day 1 (C1D1) is defined as the first day that ASTX727 is administered.

SUMMARY:
The purpose of this study is to see whether the study drug ASTX727 is an effective treatment for people who have MPNST with a PCR2 mutation.

ASTX727 is a combination of two drugs (cedazuridine and decitabine) that have been designed to target cancer cells with a PCR2 mutation and to disrupt the cells' ability to survive and grow. The study researchers think that the study drug allows decitabine to work better than decitabine given alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed PRC2 loss MPNSTs (e.g. IHC of loss H3K27me2 and/or H3K27me3 immunostaining, and/or inactivating mutations in EED, SUZ12, EZH2 by CLIA approved genetic assays), which are advanced, unresectable or metastatic and have progressed on at least one line of standard of care systemic therapy, or administration of cytotoxic chemotherapy is not considered in the best interest for the patient.
* Patients must be at least 16 years of age
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Disease must be measurable by RECIST 1.1.
* Patients must be able to take oral medications.
* Patient or legally authorized representative can understand and comply with the protocol and must sign an informed consent document.
* Adequate renal, hepatic and hematologic function as the following: serum creatinine ≤ 1.5 x upper limit of normal (ULN), total serum bilirubin ≤ 1.5 x ULN, serum AST (SGOT) ≤ 2.5 x ULN (or ≤ 5.0 x ULN if considered due to tumor (liver metastases)), serum ALT (SGPT) ≤ 2.5 x ULN (or ≤ 5.0 x ULN if considered due to tumor (liver metastases)), ANC ≥ 1500/µL, platelets ≥ 75,000/µL, and hemoglobin ≥ 9 g/dL(can be transfused to achieve this). Prothrombin time (PT), international normalized ratio (INR), and partial thromboplastin time > 1.5 x ULN. Patients on a stable maintenance regimen of anticoagulation therapy for at least 30 days prior to screening may have PT/INR measurements > 1.5 x ULN
* Patients of childbearing potential must have a negative serum pregnancy test at screening and at cycle 1 day 1 (-3 days) prior to the first dose of study therapy being administered. Female patients of childbearing potential must agree to use two reliable methods of contraception starting at signing the ICF, during and for 6 months following the last dose of study drug
* Women must agree not to breastfeed during treatment with study drug and for 2 weeks after the last dose.
* Sexually active males must agree to use a condom during intercourse and agree to not donate sperm while taking the drug and for 3 months after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men to prevent delivery of the drug via seminal fluid.

Exclusion Criteria:

* Patients have a severe and/or uncontrolled medical disease (e.g., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
* Patients have known active brain metastasis or leptomeningeal disease.
* Active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) or known active or chronic infection with human immunodeficiency virus (HIV). Prior hepatitis infection that has been treated with highly effective therapy with no evidence of residual infection (including undetectable viral loads while on antiviral therapy) and with normal liver function (ALT, AST, total and direct bilirubin ≤ ULN) is allowed.
* Known active tuberculosis.
* Concurrent active inoperable locally advanced or metastatic malignancy (except for malignancies which the treating investigator determines are unlikely to interfere with treatment and safety analysis or are less of a treatment priority than their diagnosis of advanced MPNST).
* Patients have clinically significant cardiovascular disease, including any of the following: 1) History of acute coronary syndrome including myocardial infarction, unstable angina, CABG, coronary angioplasty or stenting < 6 months prior to screening; 2) symptomatic chronic heart failure (New York Heart Association Criteria, Class II-IV); 3) evidence of clinically significant cardiac arrhythmias and/or conduction abnormalities < 6 months prior to screening except atrial fibrillation (AF) and paroxysmal supraventricular tachycardia (PSVT).
* A screening Fridericia corrected QT interval (QTcF) ≥ 450 ms (men) or ≥ 470 ms (women) (average of triplicates).
* Left ventricular ejection fraction (LVEF) <50% as determined by a multigated acquisition (MUGA) scan or echocardiogram.
* History of thromboembolic or cerebrovascular events ≤ 3 months prior to starting study treatment, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis or pulmonary emboli.
* Impairment of gastrointestinal function or gastrointestinal disease (e.g., uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, ulcerative diseases, bowel resection with decreased intestinal absorption).
* Patients had a major surgery within 3 weeks prior to study entry or who have not recovered from side effects of such procedure.
* Patients with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
* Treatment with anti-cancer therapy within 14 days prior to the first dose of study drug therapy. For prior biological therapies, e.g., monoclonal antibodies with a half-life longer than 3 days, the interval must be at least 28 days prior to the first dose of study drug.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
the best clinical benefit rate (CBR) | at the end of 16 weeks
  (complete response [CR] + partial response [PR] + stable disease [SD]) by RECIST1.1

SECONDARY OUTCOMES:
objective response rate (ORR) | 8 weeks
  by RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ping Chi, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm